CLINICAL TRIAL: NCT06359990
Title: BrotherlyACT: A Culturally Congruent and Technology-Enhanced Youth Violence and Substance Use Intervention for Black Boys and Men
Brief Title: BrotherlyACT: A Tech-Enhanced Violence and Substance Use Intervention for Black Boys and Young Men
Acronym: BrotherlyACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Chuka Emezue, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RushUMCEmezue
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Violence in Adolescence; Substance Use; Avoidance of Healthcare
Keywords: Youth violence; Substance use; Experiential avoidance; African American; Youth; Males; mHealth
MeSH Terms: conditions — Substance-Related Disorders; Treatment Refusal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrotherlyACT Intervention Group (Experimental): Three components make up BrotherlyACT: 1) Brief psychoeducational modules adapted from an evidence-based violence prevention program; 2) A Safety Planning Toolkit offering tools for risk assessment, mood tracking, goal setting, and mindfulness-based stress reduction; 3) A Service Engagement Chatbot that uses NLP to provide zip-code based navigational support and talk therapy.
  Interventions: Behavioral: BrotherlyACT
- Waitlist Control Group (WCG) (Other): Waitlist Control Group (WCG)
  Interventions: Other: BrotherlyACT Waitlist Control Group (WCG)

INTERVENTIONS:
Behavioral: BrotherlyACT — BrotherlyACT is a digital intervention to prevent youth violence and substance use among trauma-exposed young Black males, ages 125-24. This intervention combines life skills coaching, safety planning tools, and an AI-driven chatbot to reduce the risk and effects of violence and early substance use.
  Arms: BrotherlyACT Intervention Group
Other: BrotherlyACT Waitlist Control Group (WCG) — During the waiting period, participants in the control group do not receive the BrotherlyACT intervention but may continue with their usual activities or interventions.
  Arms: Waitlist Control Group (WCG)

SUMMARY:
This study will adapt and test a culturally tailored, multi-component, and trauma-focused digital intervention to reduce the risk and effects of youth violence and substance use and bridge service access gaps for young Black males (YBM) in pediatric emergency and community-based low-resource settings.

DETAILED DESCRIPTION:
Across U.S. cities, Black youth face a 20-fold higher risk, and Hispanic youth a 4.4-fold higher risk of fatal shootings compared to non-Hispanic White youth aged 18-24. Despite these disparities, young Black males (YBM) in program-rich cities report reduced service utilization and uptake due to various modifiable personal and community-based factors. Several structural discrimination and avoidance-related processes drive these factors. For instance, YBM report high levels of Service Avoidance (where YBM avoid institutions that might create official records or have law enforcement presence, fearing involvement in the judicial system). At the individual level, they also report Experiential Avoidance (where trauma-impacted YBM suppress uncomfortable thoughts, experiences, and feelings - including openness to intervention - leading to maladaptive coping strategies (e.g., retaliation and substance dependence). These issues jointly amplify youth violence (YV) risk and related issues, such as substance use (SU). Yet, few programs target these personal and structural drivers of YV and SU. The investigator's prior research involving assault-injured YBM has shown a preference for digital and remotely delivered interventions that provide personalized feedback, round-the-clock support, privacy, and integrated services. Digital interventions are an underutilized resource for helping at-risk YBMs overcome some os there personal and structural barriers to utilizing behavioral and other health services.

This research study aims to adapt, validate, and test the efficacy of BrotherlyACT, a culturally tailored, multi-component, and trauma-focused digital intervention to reduce the risk and effects of youth violence and substance use and bridge service access gaps for young Black males (YBM) in pediatric emergency and community-based low-resource settings. This study will recruit a sample of 300 assault-injured YBMs at discharge from three level 1-2 emergency departments (EDs) and violence-involved YBMs from two community-based organizations. Participants will be randomly assigned to the intervention or Waitlist Control Group (WCG). The intervention group will receive the app/web-based BrotherlyACT, comprising three main components: 1) Brief psychoeducational microlearning lesson videos based on the Acceptance and Commitment Therapy (ACT); 2) A Safety Planning Toolkit offering tools for risk assessment, emotional regulation, goal setting, and mindfulness-based stress reduction; 3) A Service Engagement Chatbot (called DEVON) that uses NLP to provide zip-code based navigational support and talk therapy. It is hypothesized that at baseline, 1-, and 3-months post-intervention, the intervention group will demonstrate reductions in 1) YV perpetration (reactive and proactive aggression); 2) YV victimization; 3) substance use (alcohol and other drug use occasions in the past 30 days, substance use attitudes and beliefs). Secondary outcomes include (A) service utilization intensity (e.g., # of weeks receiving follow-up/referral care, # of discriminatory staff-YBM encounters), (B) Experiential Avoidance, (C) Psychological distress, (D) Violence Intentions, and (E) Readiness to Change. This study will explore potential site/location and mediation/moderation effects.

ELIGIBILITY:
Inclusion Criteria:

1. Assault-injured youth without impairments (e.g., unstable injuries),
2. Male-identifying, irrespective of sexual orientation;
3. Black/African American hospitalized for injury;
4. Ages 15 to 24 years (inclusive);
5. English literate at a 5th-grade reading level or higher;
6. Able to assent/consent and provide parental consent.

Exclusion Criteria:

1. Currently detained in the criminal justice system,
2. Unable to complete assent/consent forms and assessments due to language barriers, cognitive dysfunction or injury, active psychotic disorder, suicide attempt as the mechanism of injury, and/or current treatment for depression or PTSD,
3. Those presenting with a chief complaint of acute sexual assault, suicidal ideation or attempt, or child maltreatment will be excluded as they already receive other ED services.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Males
Enrollment: 300 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
The Reactive-Proactive Aggression Questionnaire (RPQ) | Baseline, 1-, and 3-months post-intervention
  Change in the perpetration of youth and peer aggression from baseline to follow-up measured with the Reactive-Proactive Aggression Questionnaire (RPQ; Raine et al., 2006) measures two dimensions of aggression in physical or verbal forms. Scores (0, 1, or 2) for proactive aggression items (2,4,6,9,10,12,15, 17,18,20,21,23) and reactive items (1, 3, 5,7,8,11, 13,14, 16,19,22) are summated to form proactive and reactive scales. Proactive and reactive scale scores are summated to obtain total aggression scores. Higher scores obtained from the scale indicate higher levels of aggression.
Multidimensional Peer Victimization Scale (MPVS) | Baseline, 1-, and 3-months post-intervention
  Change in youth and peer violence victimization from baseline to follow-up measured with the Multidimensional Peer Victimization Scale (MPVS; Mynard & Joseph, 2000). The MPVS is a 16-item self-report instrument that contains four subscales: physical victimization, verbal victimization, social manipulation, and attacks on property. Each item is scored on a three-point Likert scale, with participants indicating how often they had experienced each of the 16 victimization experiences in the past year. Total victimization scores range from 0 to 32, with subscale scores ranging from 0 to 8. Higher scores indicate that a youth has been subjected to more incidents of peer victimization.
The Alcohol Use Disorders Identification Test (AUDIT) | Baseline, 1-, and 3-months post-intervention
  The Alcohol Use Disorders Identification Test (AUDIT) focuses on drinking patterns and alcohol-related behaviors. Research supports the use of the AUDIT for adolescents ages 14 to 18, with cut points of 2 for identifying any alcohol problem use and 3 for alcohol misuse or dependence (Knight et al., 2003). WHO recommends a total AUDIT score of ≥8 as an indicator of hazardous and harmful alcohol use, as well as possible alcohol dependence (Thomas F Babor & Robaina, 2016).
Drug Use Disorders Identification Test (DUDIT) | Baseline, 1-, and 3-months post-intervention
  Drug Use Disorders Identification Test (DUDIT) is an 11-item tool that is similar to the Alcohol Use Disorders Identification Test (AUDIT), as the DUDIT focuses specifically on drug use and consists of a series of questions designed to evaluate different aspects of drug use behavior and related consequences. As with the AUDIT, items 1 to 9 are scored on a 0 to 4 scale, with the final two questions scored 0, 2, 4. The maximum score is 44. Scoring guidelines suggest that a score of 6 or more among men and 2 or more among women may be indicative of drug-use-related problems. A score of 25 points or more, regardless of sex, strongly indicates dependence.
Change in Attitude toward Substance Use | Baseline, 1-, and 3-months post-intervention
  Increased awareness of normative beliefs and consequences related to substance use as measured by the Adolescent Attitudes Questionnaire

SECONDARY OUTCOMES:
Emotional Avoidance Strategy Inventory for Adolescents (EASI-A) | Baseline, 1-, and 3-months post-intervention
  Change in Experiential avoidance from baseline to follow-up measured using the Emotional Avoidance Strategy Inventory for Adolescents (EASI-A). The EASI-A has three subscales: Avoidance of Thoughts and Feelings, Avoidance of Emotion Expression, and Active Avoidance Coping.
The Kessler Psychological Distress Scale (K-10) | Baseline, 1-, and 3-months post-intervention
  Change in psychological distress from baseline to follow-up will be assessed using the Kessler Psychological Distress Scale (K10). Psychological Distress will be measured on a scale from five to one (5=all of the time; 4= Most of the time; 3 some of the time; 2= A little of the time; 1= none of the time). The scores range from 6 to 30, and the total scores are calculated by summing the individual items. Higher scores indicate high psychological distress.
The University of Rhode Island Change Assessment Scale (URICA) | Baseline, 1-, and 3-months post-intervention
  The University of Rhode Island Change Assessment Scale (URICA) is a 32-item self-report measure that includes four subscales measuring the stages of change or readiness to change: Precontemplation, Contemplation, Action, and Maintenance (there is also a 24-item version). Responses are given on a 5-point Likert scale ranging from (1=strong disagreement to 5=strong agreement), McConnaughy et al., 1983).
Intensity-of-Care Measurements | 3-months post-intervention
  Based on a 3-part measurement developed by the Children's Hospital of Philadelphia (CHOP) and the more standard intensity measurements of total time used by the San Francisco WrapAround care program and Healing Hurt People Program (HHP) in Philadelphia. This measurement includes 1) # of weeks receiving care, 2) # of needs addressed, and 3) # of staff-client encounters, 4) # of discriminatory staff-YBM encounters.
Violent Intentions-Teen Conflict Survey | Baseline, 1-, and 3-months post-intervention
  Measures intentions to use nonviolent strategies to control anger and conflict. These items measure intentions to use nonviolent strategies to control anger and conflict. Respondents are asked to indicate how likely they would be to adopt certain nonviolent behaviors the next time they get angry. Responses are summed' with a possible range of 8 to 32. High scores indicate a stronger intention to use non-violent strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Chuka N Emezue, PhD, MPH, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated and de-identified IPD may be made available to other scientists, policymakers, and programs/critical stakeholders working with racial and ethnic minority youth and violence prevention. Toward this end, we will create a database of all participant data, removing personal identifiers or links to participants. This database will be shared with requesters as appropriate. The purpose of the database is to enable additional exploratory analyses that may lead to additional oral presentations at scientific conferences and manuscripts. As new findings emerge from the study, we will make possible secondary analyses to explore the data further. For researchers, programs, and others who would like to use BrotherlyACT in their setting, we will work with the Rush University tech ventures office to develop a materials transfer agreement with acknowledgment of funding sources as appropriate.
Supporting Information: Study Protocol, SAP
Time Frame: As determined by funders.
Access Criteria: As described above.

REFERENCES:
- [Background] Emezue C, Karnik NS, Reeder B, Schoeny M, Layfield R, Zarling A, Julion W. A Technology-Enhanced Intervention for Violence and Substance Use Prevention Among Young Black Men: Protocol for Adaptation and Pilot Testing. JMIR Res Protoc. 2023 May 1;12:e43842. doi: 10.2196/43842. PMID 37126388
- See also: Enrolment Page — https://redcap.link/bawebsitet